CLINICAL TRIAL: NCT02133924
Title: Phase II Multicenter Study Of Natalizumab Plus Standard Steroid Treatment For High Risk Acute Graft-Versus-Host Disease
Brief Title: Multicenter Study Of Natalizumab Plus Standard Steroid Treatment For High Risk Acute Graft-Versus-Host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: John Levine (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor-Investigator, John Levine, Professor of Internal Medicine and Pediatrics, Director of BMT Clinical Research, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 15-1624
Record Dates: First submitted 2014-05-06; First posted 2014-05-08 (Estimated); Results first posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Acute Graft Versus Host Disease
Keywords: Graft vs Host Disease; Graft vs Host Reaction; allogeneic bone marrow transplantation; allogeneic hematopoietic stem cell transplantation; adverse effects
MeSH Terms: conditions — Graft vs Host Disease | interventions — Natalizumab; Steroids; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Natalizumab with steroids (Experimental): For subjects whose GVHD assay is Ann Arbor score 2 or 3, the study treatment will consist of two drugs, prednisone (or methylprednisolone) and natalizumab.
  Protocol treatment must start within 3 days of the subject's diagnosis of acute GVHD.
  Interventions: Drug: natalizumab; Drug: steroids

INTERVENTIONS:
Drug: natalizumab — Natalizumab 300mg on days 0 and 14.
  Other Names: Tysabri
Drug: steroids — Prednisone 2mg/kg/d (or methyl-prednisolone IV equivalent)
  Other Names: Prednisone; methylprednisolone equivalent IV

SUMMARY:
This research trial is designed to study the safety and effectiveness of combining the study drug, Natalizumab (Tysabri®) with the standard treatment, the use of steroids, as a new treatment for acute graft versus host disease (acute GVHD). GVHD is the most common serious complication, after bone marrow transplant. GVHD occurs when the donor cells (the graft), treat the recipient's body as "foreign" and attack the cells in the recipient's body. During this immune system response, donor cells damage body tissues, such as the skin, liver, stomach, and/or intestines. Acute GVHD can be severe and if severe, potentially fatal to the transplant recipient. Acute GVHD usually happens within the first several months after transplant.

The goal of this research is to develop a safer and more effective treatment for acute GVHD, and particularly for acute GVHD that affects the gastrointestinal (or GI) tract, with the ultimate goal being safer and more effective transplant therapies for blood cancers such as leukemia, lymphoma, and multiple myeloma.

DETAILED DESCRIPTION:
The only proven effective treatment for patients with acute graft vs host disease is steroids. Patients not responding to steroid treatment are at high risk for death. Unfortunately, based on the early symptoms, it is not possible to tell whether a patient will respond to steroids, when GVHD is diagnosed and treatment with steroids, such as prednisone, is started.

This research trial is designed to study the safety and effectiveness of combining the study drug, Natalizumab (Tysabri®) with the use of steroids to treat acute GVHD in patients at the earliest stages of clinical symptoms, but, by using a proprietary method developed at the University of Michigan and the Icahn School of Medicine at Mount Sinai, are predicted to be at high risk for not responding to steroid therapy, the standard of care.

Investigators at Mount Sinai have developed a research method believed that it might make it possible to predict who is at high risk for not responding to steroids. This method, called Ann Arbor GVHD scoring, uses the levels of naturally occurring chemicals in the blood (called biomarkers) to determine a patient's GVHD score(1, 2, or 3).

A hypothesis is that many patients with Ann Arbor score 2 or 3 GVHD, will not respond well to steroid treatment and die within 6 months of their GVHD diagnosis. Most of the deaths are due to intestinal GVHD, which sometimes does not develop, until after standard steroid treatment has already begun.

Only patients with Ann Arbor score 2 or 3 GVHD, will be eligible for this study treatment. It is important to understand that Ann Arbor GVHD grading is not approved for clinical use. It can only be used as a test for research purposes. In this study, patients must have their blood tested to determine, if they qualify as Ann Arbor score 2 or 3 GVHD, and must start the study treatment within 3 days of starting systemic steroid treatment for acute GVHD.

The study will test whether the investigators can improve steroid response and prevent death from GVHD with the combination therapy, by blocking the donor cells from getting to the intestine and causing damage. Natalizumab (Tysabri®) is a drug that works by blocking the signals that cause immune cells like donor cells, to travel to organs like the intestine or brain.

Natalizumab is FDA-approved in adults, to treat Crohn's disease, a chronic condition where immune cells cause damage to the digestive system (such as the stomach, intestines). It is also used to treat multiple sclerosis where immune cells cause damage to the nervous system in the brain. Its intended use is for patients with disease that has not responded to the standard treatment, or cannot tolerate the side effects from standard treatments.

Natalizumab has never been used for treating GVHD. It is an experimental drug for this study, because the investigators are investigating a new use for the drug, as a GVHD treatment.

ELIGIBILITY:
Inclusion Criteria:

* New onset high risk acute GVHD (Ann Arbor score 2 or3 as defined in Appendix C of the protocol) following allogeneic bone marrow transplantation. Any clinical severity (Glucksberg grade I-IV) is eligible. Patients with prior or existing diagnosis of GVHD without any treatment are eligible. Patients given only topical corticosteroids for skin GVHD are eligible.
* Any donor type (e.g., related, unrelated) or stem cell source (bone marrow, peripheral blood, cord blood). Recipients of non-myeloablative and myeloablative transplants are eligible.
* No prior systemic treatment for acute GVHD except for a maximum of 3 days of prednisone ≤2 mg/kg/day (or IV methylprednisolone). Topical skin steroid treatment, non-absorbable oral steroid treatment for GI GVHD, and resumption of GVHD prophylaxis agents (e.g., calcineurin inhibitors) are permissible. Patients enrolled in BMT CTN 1501 who randomized to sirolimus are also eligible.
* Age 18 years or older.
* Direct bilirubin must be <2 mg/dL unless the elevation is known to be due to Gilbert syndrome or aGVHD within 3 days of enrollment.
* ALT/SGPT and AST/SGOT must be <5 x the upper limit of the normal range within 3 days of enrollment, unless the elevation is due to liver GVHD.
* If the patient is a woman of child-bearing potential, the patient and their sexual partner must agree to practice effective contraception.
* Written informed consent from patient.
* Biopsy of acute GVHD target organ is strongly recommended, but not required. Enrollment should not be delayed for biopsy or pathology results. Patients who do not enroll within 3 days of systemic steroid treatment for acute GVHD are not permitted to participate.

Exclusion Criteria:

* Progressive or relapsed malignancy since BMT
* Uncontrolled active infection
* Patients with chronic GVHD only. Patient with overlap syndrome are eligible.
* History of Progressive Multifocal Leukoencephalopathy (PML)
* Known hypersensitivity to natalizumab
* Pregnant or nursing (lactating) women
* Use of other drugs for the treatment of acute GVHD
* Steroid therapy for indications other than GVHD at doses >0.5 mg/kg/d of methylprednisolone or equivalent within 7 days prior to initiation of GVHD treatment
* Patients on dialysis
* Patients requiring ventilator support
* Investigational agent within 30 days of enrollment without approval from the Sponsor-Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2021-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John E Levine, MD, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (12):
- United States (12):
  - City of Hope, Duarte, California
  - Emory University, Atlanta, Georgia
  - Northwestern, Chicago, Illinois
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinical, Rochester, Minnesota
  - Mount Sinai Health System, New York, New York
  - Columbia University, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee

REFERENCES:
- [Derived] Al Malki MM, London K, Baez J, Akahoshi Y, Hogan WJ, Etra A, Choe H, Hexner E, Langston A, Abhyankar S, Ponce DM, DeFilipp Z, Kitko CL, Adekola K, Reshef R, Ayuk F, Capellini A, Chanswangphuwana C, Eder M, Eng G, Gandhi I, Grupp S, Gleich S, Holler E, Javorniczky NR, Kasikis S, Kowalyk S, Morales G, Ozbek U, Rosler W, Spyrou N, Yanik G, Young R, Chen YB, Nakamura R, Ferrara JLM, Levine JE. Phase 2 study of natalizumab plus standard corticosteroid treatment for high-risk acute graft-versus-host disease. Blood Adv. 2023 Sep 12;7(17):5189-5198. doi: 10.1182/bloodadvances.2023009853. PMID 37235690

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment from 8/11/2016 -11/20/2020
Groups:
- Participants With High Risk Acute Graft-Versus-Host Disease: For participants whose Graft-Versus-Host Disease (GVHD) assay is Ann Arbor score 2 or 3, the study treatment will consist of two drugs, prednisone (or methylprednisolone) 2mg/kg/d (or methyl-prednisolone IV equivalent) and Natalizumab 300mg on days 0 and 14.
Period: Overall Study
Arm/Group | Participants With High Risk Acute Graft-Versus-Host Disease
Started | 76
Completed | 34
Not Completed | 42
Not completed — Death | 38
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Groups:
- Participants With High Risk Acute Graft-Versus-Host Disease: For participants whose GVHD assay is Ann Arbor score 2 or 3, the study treatment will consist of two drugs, prednisone (or methylprednisolone) 2mg/kg/d (or methyl-prednisolone IV equivalent) and Natalizumab 300mg on days 0 and 14.
Arm/Group | Participants With High Risk Acute Graft-Versus-Host Disease
Number analyzed (Participants) | 76
Age, Continuous [Median (Full Range); unit: years] | 59 [23 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 64
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 61
  More than one race | 2
  Unknown or Not Reported | 2
Diagnosis [Count of Participants; unit: Participants] — Myelodysplastic/Myeloproliferative Neoplasms (MDS/MPN)
  Chronic Myelomonocytic Leukemia (CMML)
  Chronic Lymphocytic Leukemia (CLL)
  Participants
    Acute Leukemia | 37
    MDS/MPN/CMML | 25
    Lymphoma/CLL | 8
    Multiple Myeloma | 2
    Non-Malignant | 4
Donor [Count of Participants; unit: Participants]
  Matched related | 23
  Matched unrelated | 39
  Mismatched related | 8
  Mismatched unrelated | 6
Conditioning Regimen [Count of Participants; unit: Participants] — pre-transplant conditioning regimen intensity
  Participants
    Full | 32
    Reduced | 44
Anti-thymocyte Globulin (ATG) [Count of Participants; unit: Participants]
  Yes | 7
  No | 69
GVHD Prophylaxis [Count of Participants; unit: Participants] — calcineurin inhibitor (CNI)
  mycophenolate mofetil (MMF)
  Participants
    CNI/MTX (+/- Other) | 47
    CNI/MMF (+/- Other) | 7
    CNI/sirolimus | 5
    Cyclophosphamide based | 10
    T Cell Depletion | 5
    Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response (CR)
Description: The primary endpoint for this clinical study is the proportion of complete response, CR (that is, the percent of patients with skin, liver, and GI GVHD - all stage 0) at day 28 of study treatment. Stage 0 = no rash, total bilirubin <2 mg/dl, diarrhea <500 ml/d
Time Frame: Day 28
Population: one participant data inevaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With High Risk Acute Graft-Versus-Host Disease
Number analyzed (Participants) | 75
Participants | 34

2. Secondary Outcome: Number of Participants With Overall Survival (OS)
Description: Number of participants with overall survival at 1 year
Time Frame: 1 year
Population: one participant data inevaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With High Risk Acute Graft-Versus-Host Disease
Number analyzed (Participants) | 75
Participants | 37

3. Secondary Outcome: Number of Participants With Non-Relapse Mortality (NRM)
Description: Number of participants with Non-Relapse Mortality (NRM) at 6 months and 1 year
Time Frame: 6 months and 1 year
Population: one participant data inevaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With High Risk Acute Graft-Versus-Host Disease
Number analyzed (Participants) | 75
Participants
  6 months | 25
  1 year | 28

4. Secondary Outcome: Number of Participants With SR GVHD
Description: Number of participants with steroid-refractory (SR) GVHD to express cumulative incidence of treatment-refractory GVHD (defined as absence of CR or PR on day 28 of treatment or who receive additional immunosuppression prior to day 28)
Time Frame: 1 year
Population: one participant data inevaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With High Risk Acute Graft-Versus-Host Disease
Number analyzed (Participants) | 75
Participants | 30

5. Secondary Outcome: Time to Discontinuation of Steroid Therapy
Description: Time in days to discontinuation of steroid therapy.
Time Frame: up to 365 days
Population: one participant data inevaluable
Measure: Median (Full Range); unit: days
Arm/Group | Participants With High Risk Acute Graft-Versus-Host Disease
Number analyzed (Participants) | 75
days | 108 [30 to 365]

6. Secondary Outcome: Number of Participants Who Received Additional GVHD Therapies
Description: Number of participants who received additional GVHD therapies (defined as the initiation of a new acute GVHD therapy, regardless of duration)
Time Frame: 1 year
Population: one participant data inevaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With High Risk Acute Graft-Versus-Host Disease
Number analyzed (Participants) | 75
Participants | 33

7. Secondary Outcome: Number of Serious Infections
Description: Number of serious infections (defined as score 3 by the Blood and Marrow Transplant Clinical Trials Network)
Time Frame: 6 months
Population: one participant data inevaluable
Measure: Number; unit: events
Arm/Group | Participants With High Risk Acute Graft-Versus-Host Disease
Number analyzed (Participants) | 75
events | 52

8. Secondary Outcome: Number of Participants With Overall Response Rate (CR + PR)
Description: Overall response rate (CR + PR) at day 28. Partial Response (PR) is defined as improvement in one or more organs involved with GVHD symptoms without progression in others. For a response to be scored as PR on day 28, the patient must be in PR on day 28 and have had no intervening non-study therapy for acute GVHD.
Time Frame: Day 28
Population: one participant data inevaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With High Risk Acute Graft-Versus-Host Disease
Number analyzed (Participants) | 75
Participants | 45

ADVERSE EVENTS:
Time Frame: 1 year
Description: one participant withdrew and was inevaluable for AEs
Arm/Group | Participants With High Risk Acute Graft-Versus-Host Disease
All-Cause Mortality (participants affected / at risk) | 38/75
Serious Adverse Events (participants affected / at risk) | 51/75
Other Adverse Events (participants affected / at risk) | 32/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With High Risk Acute Graft-Versus-Host Disease (N=75)
Acute Liver Injury (Hepatobiliary disorders) | 1
GVHD (Immune system disorders) | 26 — Graft Versus Host Disease
Fatigue (General disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Autonomic Disorder (Nervous system disorders) | 1
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Depression (Renal and urinary disorders) | 1
Autoimmune Encephalitis (Immune system disorders) | 1
GI Hemorrhage (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Graft Failure (Blood and lymphatic system disorders) | 1
Hemolytic Anemia (Blood and lymphatic system disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Psychosis (Psychiatric disorders) | 1
Treatment Related Secondary Malignancy (PTLD) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — PTLD: post-transplant lymphoproliferative disease
Relapse (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Thrombotic Microangiopathy (Vascular disorders) | 1
Transaminitis (Hepatobiliary disorders) | 1
Poor Graft Function (Blood and lymphatic system disorders) | 1
Sepsis (Infections and infestations) | 14
Lung Infection (Infections and infestations) | 5
Encephalitis Infection (Infections and infestations) | 3
Meningitis (Infections and infestations) | 1
Bacteremia (Infections and infestations) | 6
C. Difficile Infection (Infections and infestations) | 4
Urinary Track Infection (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Viremia (Infections and infestations) | 4
Upper Respiratory Infection (Immune system disorders) | 1
Fungemia (Infections and infestations) | 2
Duodenal Infection (Infections and infestations) | 1
EBV PTLD (Infections and infestations) | 1 — Epstein-Barr virus positive post-transplant lymphoproliferative disease
Small Intestine Infection (Infections and infestations) | 1
CNS Toxoplasmosis (Infections and infestations) | 1
Mucormycosis (Infections and infestations) | 1
Invasive fungal Infection: Aspergillus Galactomannan (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With High Risk Acute Graft-Versus-Host Disease (N=75)
Anemia (Blood and lymphatic system disorders) | 11
Anxiety (Psychiatric disorders) | 1
Hypertension (Vascular disorders) | 3
Delirium (Psychiatric disorders) | 1
Edema (General disorders) | 6
GI Hemorrhage (Gastrointestinal disorders) | 3
GVHD (Immune system disorders) | 2
Hematuria (Renal and urinary disorders) | 1
Hemolytic Anemia (Blood and lymphatic system disorders) | 1
Blood Bilirubin Increased (Investigations) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Hypotension (Vascular disorders) | 1
White Blood Cell Decreased (Investigations) | 11
Lymphocyte Count Decreased (Investigations) | 8
Neutrophil Count Decreased (Investigations) | 3
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Somnolence (Nervous system disorders) | 1
Platelet Count Decreased (Investigations) | 17
Thrombotic Microangiopathy (Vascular disorders) | 4
Fatigue (General disorders) | 5
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 3
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 1
Catheter Related Infection (Infections and infestations) | 2
Colitis (Infections and infestations) | 1
CMV Viremia (Infections and infestations) | 2
Skin Infection (Infections and infestations) | 2
Alanine Aminotransferase Increased (Investigations) | 2
Alkaline Phosphatase Increased (Investigations) | 2
Aspartate Aminotransferase Increased (Investigations) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Lung Infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/24/NCT02133924/Prot_SAP_000.pdf